CLINICAL TRIAL: NCT04856280
Title: The Effects of Kinesiological Taping and Aerobic Exercise in Women With Primary Dysmenorrhea: A Randomized Single-Blind Controlled Trial
Brief Title: Kinesiological Taping and Aerobic Exercise in Women With Primary Dysmenorrhea:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, mbudak, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KinesioExercisePD2021
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Primary Dysmenorrhea; Kinesics; Aerobic Exercise
Keywords: Primary Dysmenorrhea; Kinesiological Taping; Aerobic Exercise
MeSH Terms: conditions — Kinesics | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor was blinded regarding group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The kinesiological taping (KT) group (n=15) (Experimental): 6 sessions of taping was applied to the kinesiological taping group, starting on the 14th day of the menstrual cycle and 2 times a week for 3 weeks until the cycle ended. Using the KT ligament technique, it was applied to the supra pubic region with 100% tension in order to reduce contraction in the uterus
  Interventions: Behavioral: Kinesiological taping
- The aerobic exercise (AE) group (n=15) (Active Comparator): In the AE group, walking and climbing stairs were given during the menstrual cycle, 45 minutes session per day, 3 days a week over 3 weeks. The exercise protocol consists of 5 minute warm up, 35 min AE and 5 minute cool-down exercises. Warm-up and cool-down exercises include an active range of motion (ROM) exercises for upper and lower extremity. Aerobic exercise includes 30 min of moderate walking and climbing stairs. The aerobic exercise was performed in accordance with the definition of moderate-intensity exercise of the World Health Organization; "It was given to the participants that during moderate exercise, the individual should walk with a tempo in a way that he can speak but cannot sing"
  Interventions: Behavioral: Aerobic exercise
- The control group (n=15) (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Behavioral: Kinesiological taping — In KT Group, 6 sessions of KT were applied, starting on the 14th day of the menstrual cycle and 2 times a week for 3 weeks until the cycle ended.
  Arms: The kinesiological taping (KT) group (n=15)
Behavioral: Aerobic exercise — In the AE group, walking and climbing stairs were given during the menstrual cycle, 3 days a week, 45 minutes.
  Arms: The aerobic exercise (AE) group (n=15)

SUMMARY:
Dysmenorrhea is defined as the pain and discomfort of women during the menstrual period. Kinesiological taping (KT) and aerobic exercise (AE) are effective methods for dysmenorrhea. The purpose of this study is to investigate the effects of KT and AE on pain, attitude, depression, and quality of life in women with dysmenorrhoea. Forty-five women with dysmenorrhea wıll randomly be divided into three groups as KT group (n=15), AE group (n=15) and control group (n=15). In KT Group, 6 sessions of KT will be applied, starting on the 14th day of the menstrual cycle and 2 times per week for 3 weeks until the end of the cycle. In the AE group, walking and climbing stairs will be given during the menstrual cycle, 3 days a week, 45 minutes. No application will be applied to the control group. All groups will be evaluated with Beck Depression Scale (BDS), Mcgill Pain Questionnaire (MPQ), Menstrual Attitude Scale (MAS), and Short Form- 36 (SF-36) before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 15-30
* Not being married
* Women with abdominal pain during menstruation 5 and above according to the Visual Analogue Scale.
* Women whose menstrual cycle has started and those whose cycle continues.

Exclusion Criteria:

* Endometriosis and adenomyosis
* Myoma
* Endometrial polyp
* Previous pelvic infections
* Intrauterine device use
* Venous congestion in the internal genital organs

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — healthy young women who have primary dysmenorrhoea
Enrollment: 45 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Mcgill Pain Questionnaire | 4 weeks
  This questionnaire consists of 11 words to determine the sensory state of pain, and 15 words related to the quality of pain in total, consisting of 4 different words to determine its affective aspect. In addition, the pain intensity felt during measurement is measured by Visual analog Scale (VAS), and the total pain intensity assessed is measured by a 6-point Likert-type scale. In this scale, "0" is defined as no pain, "5" is defined as unbearable pain.
Menstrual Attitude Scale | 4 weeks
  The scale was prepared based on the theory that there may be versatility in menstrual attitudes, positive attitudes may occur as well as negative, and expectations that may occur according to physiological and emotional symptoms before or during menstruation may be effective in the behaviors shown in this period. Menstrual Attitude Scale (MAS) contains 33 items to measure the positive and negative attitudes of menstruation. MAS has 5 subscales such as the menstruation as a weakening phenomenon (12 no pain, unbearable pain, 32 items), the menstruation as a disturbing phenomenon (6 items), the menstruation as a natural phenomenon (5 items), the predicting/sensing that there will be menstruation (5 items), and the denying the effects of menstruation (7 items). The scale is of 5-point Likert type. The high average score of the subscales shows that the attitude towards menstruation is "positive"

SECONDARY OUTCOMES:
Beck Depression Scale | 4 weeks
  It is a test containing 21 items that the person evaluates himself. It measures the symptoms seen in depression such as emotional, cognitive and motivational. The items determine a behavioral feature related to depression. Items are numbered from 0 to 3. The goal is to objectively break down the degree of symptoms.
  The total score of all answers is calculated as follows:
  * 0 to 9 points: Minimally depressive symptoms
  * 10 to 16 points: Mild depressive symptoms
  * Between 17 and 29 points: Moderate depressive symptoms
  * Between 30 and 63 points: Severe depressive symptoms
Short Form- 36 | 4 weeks
  Short Form- 36 (SF-36) is a 36-question self-assessment scale consisting of eight subscales. This scale is based on physical function (10 items), role limitations due to physical (4 items) and emotional problems (3 items), pain (2 items), vitality (4 items), social function (2 items), mental health (5 items) and general health (5 items) subscales. Each subscale is scored between 0-100 and "0" indicates the lowest and "100" shows the best quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Miray BUDAK, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data not available due to ethical issues